CLINICAL TRIAL: NCT04413058
Title: Menstrual Cycle Characteristics of Healthcare Professionals at Covid 19 Pandemic Hospital
Brief Title: Menstrual Cycle Characteristics of Healthcare Professionals
Status: Completed | Type: Observational
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sevcan Arzu Arinkan, Medical Doctor, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: HNEAH KAEK 2020/KK/; Ministry of Health (Registry Identifier: Sevcan Arzu ARINKAN-2020-05-03T22_54_16)
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-05

CONDITIONS: Menstrual Irregularity; Covid 19
Keywords: health care professionals; menstrual cycle; Covid 19; Pandemia
MeSH Terms: conditions — Menstruation Disturbances; COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female healthcare workers: Healthy female healthcare workers at Covid 19 clinic in Istanbul, Turkey

SUMMARY:
The Covid-19 pandemic has impacted healthcare workers physically and psychologically. The aim of this study is to examine whether there is a change in menstrual cycle characteristics during pandemia. The aim of this study is to investigate whether there is an association between covid infection and menstrual cycle changes.

DETAILED DESCRIPTION:
The Covid-19 pandemic has impacted healthcare workers physically and psychologically. Healthcare workers have ben required to work under stressful conditions and take difficult decisions involving ethical implications. Increasing work demands on healthcare professionals conflict with their duties to family and friends, which causes psychological stress. All of these factors may negatively affect their menstrual cycle.

The aim of this study is to examine whether there is a change in menstrual cycle characteristics during pandemia. Second aim is to investigate whether there is an association between Covid 19 infection and menstrual cycle changes.

This cross-sectional study is conducted with healthy female participants who are working at Haydarpasa Numune Research and Training Hospital in Turkey. The researcher investigates the characteristics of menstrual cycle in female healthy workers employed in Covid 19 pandemic inpatient and outpatient clinics. The participants who are sure about their pertinent information are enrolled in the study. The exclusion criteria includes pregnancy, history of hysterectomy, oophorectomy, diseases like Asherman's syndrome and also history of endocrine disorders (progesterone deficiency, thyroid disorders and diabetes mellitus), oral contraceptive use, malignancy, primary amenorrhea, menopause and lactation.

After informed consent, detailed information is collected using structured questionnaires about their reproductive factors and menstrual cycles by direct interviews. The questionnaire contains questions about age, work experience, marital status, height, weight, working hours, use of medication, menstrual cycle characteristics (including cycle duration, duration and amount of bleeding, bleeding during the cycle, regular or irregular menstrual cycles) and dysmenorrhea. Also, the difference in menstrual cycle characteristics between covid positive and negative healthcare professionals is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Working at Covid 19 Pandemic Hospital
* Being at between 18 and 47 years old
* Having menstruation

Exclusion Criteria:

* Oral contraceptive users
* Pregnants
* Having malignancy
* Having primary amenorrhea
* Being at menopause
* Lactation

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy female healthcare workers at Covid 19 pandemic hospital
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Rate of irregular menstrual cycle | 1 month after starting to work at pandemic clinic
  Irregular menstrual cycle
Length of cycle | 1 month after starting to work at pandemic clinic
  Length of cycle (day)
Rate of prolonged bleeding | 1 month after starting to work at pandemic clinic
  Duration of bleeding (day)
Amount of flow | 1 month after starting to work at pandemic clinic
  Number of used tampons during bleeding
Rate of dysmenorrhea | 1 month after starting to work at pandemic clinic
  Dysmenorrhea status

SECONDARY OUTCOMES:
The number of difference in menstrual cycle length | Up to 1 month after covid infection
  Menstrual cycle difference between covid positive and negative healthcare workers (days)
The number of difference in bleeding days | Up to 1 month after covid infection
  Duration of bleeding difference between covid positive and negative healthcare workers (days)
The number of difference in amount of flow | Up to 1 month after covid infection
  Amount of flow difference between covid positive and negative healthcare workers (tampons)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Attarchi M, Darkhi H, Khodarahmian M, Dolati M, Kashanian M, Ghaffari M, Mirzamohammadi E, Mohammadi S. Characteristics of menstrual cycle in shift workers. Glob J Health Sci. 2013 Feb 28;5(3):163-72. doi: 10.5539/gjhs.v5n3p163. PMID 23618486
- [Background] Moen BE, Baste V, Morken T, Alsaker K, Pallesen S, Bjorvatn B. Menstrual characteristics and night work among nurses. Ind Health. 2015;53(4):354-60. doi: 10.2486/indhealth.2014-0214. Epub 2015 Apr 24. PMID 25914071
- [Background] Ok G, Ahn J, Lee W. Association between irregular menstrual cycles and occupational characteristics among female workers in Korea. Maturitas. 2019 Nov;129:62-67. doi: 10.1016/j.maturitas.2019.07.019. Epub 2019 Aug 2. PMID 31547916
- [Background] Wan GH, Chung FF. Working conditions associated with ovarian cycle in a medical center nurses: a Taiwan study. Jpn J Nurs Sci. 2012 Jun;9(1):112-8. doi: 10.1111/j.1742-7924.2011.00191.x. Epub 2011 Sep 16. PMID 22583945

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT04413058/Prot_SAP_000.pdf